CLINICAL TRIAL: NCT05785845
Title: A Phase I Trial of Computed Tomography-Guided Stereotactic Adaptive Radiotherapy (CT-STAR) for the Treatment of Central and Ultra-Central Early-Stage Non-Small Cell Lung Cancer
Brief Title: Computed Tomography-Guided Stereotactic Adaptive Radiotherapy (CT-STAR) for the Treatment of Central and Ultra-Central Early-Stage Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202302003
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Early Stage Non-small Cell Lung Cancer; Non-small Cell Lung Cancer
Keywords: NSCLC; lung cancer; ultra-central lung cancer; SBRT; IGRT; adaptive radiotherapy; CT-guided radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Computed Tomography-Guided Stereotactic Adaptive Radiotherapy (CT-STAR) (Experimental): In this study, consenting and eligible patients will receive a prescription dose of 55 Gy in 5 fractions (when possible) delivered on consecutive business days with adaptation based on daily anatomic changes as per clinical standard of care.
  Interventions: Radiation: Computed tomography-guided stereotactic adaptive radiotherapy; Device: ETHOS

INTERVENTIONS:
Radiation: Computed tomography-guided stereotactic adaptive radiotherapy — Fractions will be delivered on consecutive business days.
  Other Names: CT-STAR
Device: ETHOS — ETHOS is a unique ring-gantry CT-guided linear accelerator notable for having an on-board cone beam CT (CBCT) imaging unit with improved definition and resolution to enable target and organ-at-risk contouring. It also has a dedicated artificial intelligence treatment planning system to allow for online adaptive radiotherapy.

SUMMARY:
This study will evaluate the impact of CT-guided adaptive stereotactic radiotherapy (CT-STAR) to central and ultra-central early-stage non-small cell lung cancers on grade 3 or greater toxicity. Online adaptive radiation therapy was until recently only done clinically on an integrated MRI-guided system, but recently, Varian Medical Systems has created a CT-guided radiotherapy machine capable of online adaptive radiotherapy (ETHOS). The vast majority of stereotactic body radiotherapy (SBRT) for early-stage lung cancers is performed on a CT-guided machine rather than an MRI-guided machine, necessitating the evaluation of adaptive radiotherapy using ETHOS in this population. Historically, the non-adaptive, stereotactic treatment of central and ultra-central thoracic disease has been associated with unacceptable rates of grade 3+ toxicity. This has resulted in widespread adoption of a hypofractionated, less ablative 8-15 day treatment courses, with a baseline, one-year grade 3+ toxicity rate of 20%. Use of CT-STAR with daily, CT-guided plan adaptation to carefully spare adjacent organs-at-risk (OAR) in this setting may enable safe delivery of a shorter (5 fraction) and more ablative radiotherapy course.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiographically diagnosed stage I-IIA (AJCC, 8th ed.) non-small cell lung cancer or mediastinal recurrent non-small cell lung cancer with plans to be treated with definitive intent SBRT alone.

  * Clinical AJCC stage I defined as stage 1A1 (T1a1N0M0, T1a tumor less than or equal to 1 cm), stage 1A2 (T1bN0M0, T1b tumor between 1 and 2 cm), and stage 1A3 (T1cN0M0, T1c tumor between 2 and 3 cm).
  * Clinical AJCC stage IB defined as T2aN0M0, T2a tumor between 3 and 4 cm.
  * Clinical AJCC stage IIA defined as T2bN0M0, T2b tumor between 4 and 5 cm.
* Lesions must be defined as central or ultra-central according to the Hilus-trial13 criteria:

  * Central lesions are defined as lesions 1 cm or less from the trachea, carina, main bronchi, bronchus intermedius, or lobar bronchi.
  * Ultra-central lesions are defined as lesions touching the trachea, carina, main bronchi, bronchus intermedius, or lobar bronchi. Lesions that touch the esophagus, great vessels, or heart may also be included as ultra-central.
* Tumor coverage is deemed adequate in simulation treatment planning as determined by the treating and study physicians. Specifically, the dose to 98% of the GTV must be greater than 45 Gy.

  * Note: patients with inadequate tumor coverage at simulation will be considered screen-failures and treated off-protocol as per institutional standard-of-care. *In a in silico analysis of these patients, only 1/6 patients screen-failed based on this inclusion criteria.
* Patients should be able to hold their breath for 10 seconds.
* Inoperable disease or patient has refused/declined surgery.
* Deemed medically fit for SBRT by the treating physician.
* At least 18 years of age.
* Zubrod Performance Status 0-2 within 30 days prior to registration.
* Appropriate stage for protocol entry based upon the following minimum diagnostic workup.

  * History/physical examination within 30 days prior to registration.
  * FDG-PET/CT scan and/or CT chest (with or without contrast) for staging within 60 days prior to registration.
* Adequate bone marrow and hemostasis function determined no more than 30 days prior to registration, defined as follows:

  * Platelets ≥ 150,000 cells/mm3
  * Hemoglobin ≥ 8 g/dl
* Able to understand and willing to sign an IRB approved written informed consent.

Exclusion Criteria:

* Lesions appearing to extend through the bronchial or great vessel walls on CT imaging.
* Prior or concurrent malignancies, unless the natural history of the prior or concurrent malignancy does not have the potential to interfere with the interpretation of the results of the study.
* Patients with a pre-existing, active diagnosis of metastatic cancer.
* Severe, active comorbidity, defined as follows:

  * Unstable angina, history of myocardial infarction and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
* Past history of radiotherapy within the projected treatment field of any of the disease sites to be treated by CT-guided SBRT.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of the start of SBRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3 or greater treatment-related toxicity | 12 months post-completion of treatment (estimated to be 12 months and 5 days)
  -Toxicity graded per CTCAE version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Samson, M.D., MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu